CLINICAL TRIAL: NCT05716425
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Study Evaluating the Efficacy and Safety of STI-1558 in Adult Subjects With Mild or Moderate (COVID-19)
Brief Title: Study to Assess the Efficacy and Safety of STI-1558 in Adult Subjects With Mild or Moderate (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang ACEA Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPR-COV-301CN
Record Dates: First submitted 2023-02-03; First posted 2023-02-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — STI-1558

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): * STI-1558
  * n=600
  Interventions: Drug: STI-1558
- Arm B (Placebo Comparator): * Placebo
  * n=600
  Interventions: Drug: STI-1558 placebo

INTERVENTIONS:
Drug: STI-1558 — STI-1558 will be orally administered under fasting condition twice daily (BID) for 5 days (10 doses in total) at a dose of 600 mg, respectively; the two doses administered will be at a minimum interval of 8 hours (≥8 h). Efficacy and safety will be assessed until D29 after the first dose.
  Arms: Arm A
Drug: STI-1558 placebo — STI-1558 placebo will be orally administered under fasting condition twice daily (BID) for 5 days (10 doses in total) at a dose of 0 mg, respectively; the two doses administered will be at a minimum interval of 8 hours (≥8 h). Efficacy and safety will be assessed until D29 after the first dose.
  Arms: Arm B

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study to evaluate the efficacy and safety of STI-1558 in adult subjects with mild/moderate COVID-19. One thousand and two hundred adult subjects with mild/moderate COVID-19 (including subjects with high risk factors for progression into severe cases) are planned to be enrolled and randomized in a ratio of 1:1 into the test group or the placebo group (600 in the test group and 600 in the placebo group).

DETAILED DESCRIPTION:
One thousand and two hundred adult subjects with mild/moderate COVID-19 (including subjects with high risk factors for progression into severe cases) are planned to be enrolled and randomized in a ratio of 1:1 into the test group or the placebo group. Randomization and stratification factors include clinical type (mild vs. moderate) of COVID-19, high risk factors for severe disease (with vs. without), history of SARS-CoV-2 vaccination or infection (yes vs. no). Subjects in the test group will receive STI-1558, and subjects in the placebo group will receive STI-1558 placebo. STI-1558 and STI-1558 placebo will be orally administered under fasting condition twice daily (BID) for 5 days (10 doses in total) at a dose of 600 mg and 0 mg, respectively; the two doses administered will be at a minimum interval of 8 hours (≥8 h). Efficacy and safety will be assessed until D29 after the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥18 years;
2. Subjects comply with the diagnostic criteria for mild or moderate COVID-19 specified in the Protocol for the Diagnosis and Treatment of Novel Coronavirus Pneumonia (Trial Version 9) released by China's National Health Commission;
3. First presence of positive RT-PCR or rapid antigen assay for SARS-CoV-2 with nasopharyngeal or oropharyngeal swabs within 4 days prior to the first dose (≤4 days from the first dose);
4. First presence of at least 1 of 14 symptoms of COVID-19 within 3 days prior to the first dose (≤3 days/72 hours from the first dose) ;
5. Subjects with at least 2 of 11 target symptoms of COVID-19 within 24 hours prior to the first dose (≤24 hours from the first dose), including at least 1 designated symptom (Stuffy or runny nose, Sore throat or dry throat, Cough, Feeling hot or feverish, Shortness of breath or difficulty breathing), and score of at least 1 designated symptom ≥2 ;
6. Women of childbearing potential (WOCBP) (women of non-childbearing potential defined as women who have undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy or bilateral tubal ligation/closure, or who are infertile due to a congenital or acquired condition, or sexually mature women spontaneously menopausal for ≥ 12 months) must have a negative pregnancy test during the screening period;
7. Female subjects of childbearing potential or male subjects whose partners are of childbearing potential must agree to use a highly effective contraceptive method from screening to 30 days after the last dose;
8. Can understand and abide by the procedures and methods of this clinical trial.

Exclusion Criteria:

1. Known allergy to any ingredient of the study drug;
2. Subjects comply with the diagnostic criteria for severe or critical COVID-19 specified in the Protocol for the Diagnosis and Treatment of Novel Coronavirus Pneumonia (Trial Version 9) released by China's National Health Commission prior to the first dose;
3. Subjects urgently require or is expected to require nasal high-flow oxygen therapy or non-invasive positive pressure ventilation, invasive mechanical ventilation or ECMO prior to the first dose;
4. Subjects with abnormal liver function at screening: total bilirubin ≥ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 × ULN;
5. Subjects with active or uncontrolled hepatopathy: including cirrhosis, Child-Pugh grade B or C, acute liver failure, etc.;
6. Subjects with concomitant severe renal insufficiency (estimated glomerular filtration rate [eGFR]<45 mL/min, calculated using the serum creatinine based Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation, refer to Appendix 6 for the calculation formula) or on continuous renal replacement therapy, hemodialysis or peritoneal dialysis;
7. Subjects with impaired immune system (including subjects who are on systemic or inhaled corticosteroids or other immunosuppressants, or subjects with cancer progression or recurrence, or with human immunodeficiency virus [HIV] infection);
8. Subjects with acute episodes of chronic respiratory diseases (including bronchial asthma, chronic obstructive pulmonary disease, etc.);
9. Subjects with a history of dysphagia or any gastrointestinal disorder that affects drug adsorption;
10. Subjects with suspected or confirmed acute systemic infections other than COVID-19 (e.g., concomitant influenza), which may interfere with the evaluation of responses to the study intervention;
11. Subjects who have underwent major surgery within 14 days prior to the first dose, or have not completely recovered from surgery or plan to undergo surgery during the study period;
12. Subjects with complications that are, in the opinion of the investigator, life-threatening within 30 days prior to the first dose;
13. Subjects have received anti-SARS-CoV-2 chemical drugs such as 3CL protease inhibitors or RNA dependent RNA polymerase (RdRp) inhibitors or angiotensin converting enzyme 2 (ACE-2) and transmembrane protease serine 2 (TMPRSS2) degrading agents within 14 days prior to the first dose;
14. Subjects have received COVID-19 patients' convalescent plasma or COVID-19 human immunoglobulin or interleukin-6 (IL-6) inhibitors or anti-SARS CoV-2 neutralizing antibodies within 30 days or 5 half-lives (whichever is longer) prior to the first dose;
15. Subjects have had any SARS-CoV-2 vaccination within 3 months prior to the first dose;
16. Subjects have received any potent inhibitor or inducer of cytochrome P450 (CYP) 3A4 within 28 days or 5 half-lives (whichever is shorter) prior to the first dose;
17. Subjects who are currently participating in an interventional clinical study of other investigational drugs or devices, including other studies on COVID-19;
18. Subjects have received any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the first dose;
19. Subjects have previously participated in this study or other studies of STI-1558;
20. Pregnant or lactating women;
21. Subjects with active serious mental illness, medical disorder or other symptoms/conditions that, in the opinion of the investigator, may affect treatment, compliance or the ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1218 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Time from the first dose to sustained recovery from 11 target symptoms of COVID-19. | Time from the first dose to the day when the score of each of the 11 target symptoms of COVID-19 is 0.
  Sustained recovery from 11 target symptoms of COVID-19: the score of each of the 11 target symptoms of COVID-19 in the subject is 0 for ≥2 days.

SECONDARY OUTCOMES:
Change from baseline in the SARS-CoV-2 RNA load (reverse transcriptase polymerase chain reaction [RT-PCR] assay) at each visit point from the first dose to Day4 and Day6. | From the first dose to Day4 and Day6.
  Change from baseline in the SARS-CoV-2 RNA load at each visit point.
Time from the first dose to sustained recovery from 5 designated symptoms of COVID-19. | Time from the first dose to the day when the score of each of the 5 designated symptoms of COVID-19 is 0.
  Sustained recovery from 5 designated symptoms of COVID-19: the score of each of the 5 designated symptoms of COVID-19 (fever or feeling hot, cough, nasal obstruction or rhinorrhoea, pain pharynx or dry throat, shortness of breath or dyspnea) in the subject is 0 for ≥2 days.
Proportion of subjects with negative SARS-CoV-2 RNA conversion at each visit from the first dose to Day14. | From the first dose to Day14.
  Proportion of subjects with negative SARS-CoV-2 RNA conversion at each visit.
Area under the SARS-CoV-2 RNA load-time curve (AUC) between the first dose and Day6. | From the first dose to Day6.
  Area under the SARS-CoV-2 RNA load-time curve (AUC) .
1.Time from the first dose to sustained remission of 11 target symptoms of COVID-19. 2.Time from the first dose to sustained remission of 5 designated symptoms of COVID-19. 3.Time from the first dose to sustained remission of 14 symptoms of COVID-19. | From the first dose to the day when the score of each of the COVID-19 symptoms is 0 or 1.
  Sustained remission of the symptoms of COVID-19: the score of each of the symptoms of COVID-19 in the subject is 0 or 1 for ≥2 days; time from the first dose to sustained remission of the symptoms of COVID-19: time from the first dose to the day when the score of each of the symptoms of COVID-19 is 0 or 1.
1.Time to sustained recovery/sustained remission. 2.Proportion of subjects with sustained recovery/sustained remission. 3.Proportion of each of 11 target symptoms by severity. 4.Scores of 11 target symptoms -time AUC from the first dose to Day14. | From the first dose to Day29/Day14.
  1. Sustained recovery from 11 target symptoms of COVID-19: the score of each of the 11 target symptoms of COVID-19 in the subject is 0 for ≥2 days; time from the first dose to sustained recovery from 11 target symptoms of COVID-19: time from the first dose to the day when the score of each of the 11 target symptoms of COVID-19 is 0.
  2. Sustained remission of 11 target symptoms of COVID-19: the score of each of the 11 target symptoms of COVID-19 in the subject is 0 or 1 for ≥2 days; time from the first dose to sustained remission of 11 target symptoms of COVID-19: time from the first dose to the day when the score of each of the 11 target symptoms of COVID-19 is 0 or 1.
Proportion of subjects: 1.Progressing into severe COVID-19. 2.Undergoing COVID-19 associated hospitalization or all-cause deaths. 3.Requiring assisted oxygen inhalation/ mechanical ventilation/ECMO. 4.Admitted into the ICU. 5.Number of days in ICU. | From the first dose to Day29.
  Proportion of subjects progressing into severe COVID-19/undergoing COVID-19 associated hospitalization or all-cause deaths/requiring assisted oxygen inhalation/admitted into the intensive care unit (ICU) / requiring mechanical ventilation/extracorporeal membrane oxygenation.
During treatment: 1. Incidence of all adverse events (AEs) and serious adverse events (SAEs); 2. Any clinically significant abnormality in vital signs or physical examination; 3. Any clinically significant abnormality in laboratory tests, ECG, etc. | From the signing of informed consent to the 29 th day of administration.
  Incidence of all AEs and SAEs;Any clinically significant abnormality in vital signs or physical examination or laboratory tests, ECG, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Shenzhen Third People 's Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang R, Han B, Xu W, Zhang X, Peng C, Dang Q, Sun W, Lin L, Lin Y, Fan L, Lv D, Shao L, Chen Y, Qiu Y, Han L, Kong W, Li G, Wang K, Peng J, Lin B, Tong Z, Lu X, Wang L, Gao F, Feng J, Li Y, Ma X, Wang J, Wang S, Shen W, Wang C, Yan K, Lin Z, Jin C, Mao L, Liu J, Kushnareva Y, Kotoi O, Zhu Z, Royal M, Brunswick M, Ji H, Xu X, Lu H. Olgotrelvir as a Single-Agent Treatment of Nonhospitalized Patients with Covid-19. NEJM Evid. 2024 Jun;3(6):EVIDoa2400026. doi: 10.1056/EVIDoa2400026. Epub 2024 May 28. PMID 38804790